CLINICAL TRIAL: NCT03452059
Title: Prospective, Multicenter, Self Controlled Evaluation of the Effectiveness and Safety of Lower Limb Exoskeleton Rehabilitation Training Robot
Brief Title: Evaluation of the Effectiveness and Safety of AI-Robotics
Acronym: ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AI-Robotics Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ART-1
Record Dates: First submitted 2017-05-23; First posted 2018-03-02 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Lower Extremity Motor Dysfunction, Spinal Cord Injury
Keywords: Paralysis; Lower Extremities; Ai-Robotics
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AiLegs/AiWalker (Experimental): use of lower extremity rehabilitation training robot assisted walking (including AiLegs, AiWalker)
  Interventions: Device: AiLegs, AiWalker and HKAFO
- HKAFO/RGO (Active Comparator): use hip and knee ankle foot orthosis (HKAFO) assisted walking
  Interventions: Device: AiLegs, AiWalker and HKAFO

INTERVENTIONS:
Device: AiLegs, AiWalker and HKAFO — 5 days. Using their own control method, each morning using AiLegs, AiWalker AiWalker and HKAFO for 6 minutes walk test, three kinds of appliance between at least 30 minutes to determine heart rate, blood pressure and breathing back to quiet level. Repeat the same procedure in the afternoon ，the order is also random. Each participant will complete 10 groups of lower limb exoskeleton rehabilitation Training robot (including AiLegs, AiWalker two models) and HKAFO 6 minutes walking test

SUMMARY:
Evaluation of the effectiveness and safety of the lower extremity exoskeleton rehabilitation training robot

DETAILED DESCRIPTION:
Evaluation of the effectiveness and safety of the lower extremity exoskeleton rehabilitation training robot developed by AI-Robotics Technology Co., Ltd., Beijing for who had lower limb paralysis

ELIGIBILITY:
Inclusion Criteria:

1. more than18 but less than 60 years old，less than 80 kilos of weight，Gender is not limited
2. Confirmed by MR/CT，AIS spinal cord injury grade: A-C level (without walking ability)：Damage plane T6-L2
3. The muscle tension of the modified Ashworth grade level is less than or equal to 2
4. The range of passive motion of the hip and knee joint of the patient is approximately normal in the ankle joint Neutral position
5. Upper limb strength and physical strength are sufficient to stabilize the crutches
6. Patients are able to understand and actively participate in the training program, agree and sign the informed consent form

Exclusion Criteria:

1. The range of motion of the joints is severely limited and the walking action is limited
2. Spinal fractures are not completely healed, the clinical situation is unstable; if not fully confirmed,please go department of orthopedics or other clinical departments for diagnosing
3. Skin injury or infection of the lower extremities or the part of wearing robot
4. Unstable angina, severe arrhythmia and other heart diseases
5. Severe chronic obstructive pulmonary disease
6. Unilateral neglect
7. Severe cognitive or visual impairment
8. Other contraindications or complications that may affect walking training
9. Pregnant or lactating women
10. The investigators find that patients with poor compliance, unable to complete the study in accordance with the requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-01-13 (Actual); Study Completion 2018-01-13 (Actual)

PRIMARY OUTCOMES:
Walking efficiency | 6 minute
  6 minute walk distance,measured by meters
Walking efficiency | 6 minute
  average heart increasing rate,measured by times/min

SECONDARY OUTCOMES:
Cardiovascular response | during 6 minute walk test and right before the 6MWT
  heart rate during and after 6 minute walk test
efficiency of put on or take off the Ailegs/Aiwalker/HKAFO | immediately before beginning (pre-) and immediately after finishing (post-) each of 6 minute walk test
  to measure the time of putting on or taking off the Ailegs/Aiwalker/HKAFO before or after 6 min walk test
RPE questionaire | after 6 minute walk test
  the RPE is recorded after the 6 min walk test

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No